CLINICAL TRIAL: NCT05905315
Title: Primary Chemoradiation VS. Neoadjuvant Chemotherapy Followed By Surgery As Treatment Strategy For Locally Advanced Vulvar Carcinoma
Brief Title: Primary Chemoradiation VS. Neoadjuvant Chemotherapy Followed By Surgery As Treatment Strategy For LAVC
Acronym: VULCANIZE-II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22VL2
Record Dates: First submitted 2022-12-12; First posted 2023-06-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Vulvar Carcinoma; Squamous Cell Carcinoma of the Vulva
MeSH Terms: interventions — Paclitaxel; Carboplatin; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary chemoradiation (Active Comparator): Patients included in the standard treatment arm will receive a combination of weekly cisplatin combined with 30 fractions of external beam radiotherapy on the primary tumour with a total dose of 64.5 Gy. Cisplatin will be given for six weeks intravenously with a dose of 40 mg/m2, if possible on the first day of the week. On day 1 until day 5 the patient will receive external beam radiotherapy. This will be repeated for a six-week period.
  Interventions: Combination Product: Chemoradiation
- NACT (3-weekly carboplatin and paclitaxel) followed by surgery (Experimental): Patients included in the experimental arm will be treated with intravenous infusion of paclitaxel 175 mg/m2, followed by carboplatin 5 area under the curve (AUC). This will be administered in a 3-weekly scheme with preferably 3 and a maximum of 4 courses, with evaluation after two courses of chemotherapy by physical examination. NACT will be subsequently followed by radical surgery in responding patients. A four to six weeks interval after the last course of chemotherapy needs to be respected before surgery, to allow sufficient physical recovery.
  Interventions: Drug: Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: Paclitaxel and Carboplatin — Paclitaxel 175 mg/m2, followed by carboplatin 5 area under the curve (AUC). This will be administered in a 3-weekly scheme.
  Arms: NACT (3-weekly carboplatin and paclitaxel) followed by surgery
Combination Product: Chemoradiation — According to standard treatment.
  Arms: Primary chemoradiation

SUMMARY:
A phase 2 randomised controlled trial will be performed in which the efficacy and safety of standard treatment (primary chemoradiation; consisting of 64.5 Gy in 30 fractions of external beam radiotherapy with weekly cisplatin for six weeks) and experimental treatment (NACT; consisting of carboplatin and paclitaxel in a 3-weekly scheme) will be compared in 98 patients with LAVC, registered from eight national medical centres.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years
* Signed and written informed consent.
* Histologically-confirmed primary or recurrent squamous cell carcinoma vulvar cancer FIGO stage Ib - IVa, T1b or higher, any N, M0.
* Local tumour through which the size or localization implies requirement of treatment through primary chemoradiation or surgery consisting of extensive surgery (meaning surgery damaging pelvic organs or exenterative surgery). This can imply;

  * T1b or larger tumour with (irresectable) groin metastases
  * T1b or larger tumour with a close relationship to and/or involvement of the urethra or anal sphincter
* World Health Organization performance status of 0-2
* Adequate haematological function defined by platelet count >100x10E9/L, absolute leukocyte >3X10E9/L or neutrophil count (ANC) >1.5x10E9/L, and hemoglobin >6.0 mmol/L
* Adequate hepatic function defined by a total bilirubin level ≤1.5x the upper limit of normal (ULN) range and ASAT and ALAT levels ≤2.5x ULN for all subjects
* Adequate renal function defined by an estimated creatinine clearance ≥50mL/min according to the Cockroft-Gault formula (or local institutional standard method)
* Beta HCG level of 14 mIU/mL or below for women of childbearing potential
* Highly effective contraception for patients if the risk of conception exists

Exclusion Criteria:

* Patients with highly suspicious or positive metastases to the pelvic lymph nodes

  * Patients eligible for radical local excision without involvement of other organs
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Prior radiotherapy to the pelvis or groin area limiting full dose chemoradiation according to protocol
* Existing neuropathy which will hinder the intake of chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Vulva carcinoma
Enrollment: 98 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Loco-regional control after 24 months per completed treatment including salvage treatment | 24 months after completed treatment
  Proportion of patients free from local-regional progression

SECONDARY OUTCOMES:
Disease-related treatment failure | 24 months after completed treatment
  Patients without an event will be censored at their last date of contact. The Kaplan-Meier method will be used to estimate freedom from disease-related failure. Difference between the two main treatment arms, NACT vs. chemotherapy, will be tested using a log-rank test. Incidences of disease-related failure will be reported based on the Kaplan-Meier estimates, together with confidence intervals for the hazard ratio using both 90 and 95% confidence levels.
Disease free survival | 24 months after completed treatment
Patterns of recurrence of disease | 24 months after completed treatment
  Type of recurrence after treatment: local, regional or distant recurrence
Overall survival | 24 months after completed treatment
Treatment related death | 24 months after completed treatment
Prevention of trimodal treatment | 24 months after completed treatment
  Proportion of patients that don't need adjuvant surgery (arm 1) and number of patients that don't need adjuvant radiotherapy (arm 2)
Functional organ preservation | 24 months after completed treatment
  Proportion of patients for who an organ-sparing surgery is possible
Short term and long term complications | 24 months after completed treatment
  According to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Amant, Prof., Principal Investigator — NKI-AvL
Locations (2):
- Netherlands (2):
  - NKI-AVL, Amsterdam
  - LUMC, Leiden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amant F, van Velzen AF, Reyners A, Zijlmans H, Schaake EE, Nooij L. Primary chemoradiation versus neoadjuvant chemotherapy followed by surgery as treatment strategy for locally advanced vulvar carcinoma (VULCANize2). Int J Gynecol Cancer. 2024 Oct 7;34(10):1639-1642. doi: 10.1136/ijgc-2024-005493. PMID 38719277